CLINICAL TRIAL: NCT05732714
Title: Long Term Cardiovascular Disease Event Risk for Patients Undergoing Major Non-Cardiac
Brief Title: Long Term Cardiovascular Disease Event Risk for Patients Undergoing Major Non-Cardiac Surgery
Acronym: CVD-10y-postop
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5869
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases; Risk Reduction Behavior
Keywords: Intermediate to high risk non-cardiac surgery
MeSH Terms: conditions — Cardiovascular Diseases; Risk Reduction Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Healthy lifestyle behaviors around the time of surgery — Healthy lifestyle choices, such as improving diet and beginning to exercise around the time of surgery and it's influence on an individual's long term risk of developing cardiovascular disease.

SUMMARY:
The goal of this observational study is to learn whether the healthy lifestyle choices made around surgery can influence an individual's long term risk of developing cardiovascular disease. Patients will be observed 1-month prior to and 3-months following surgery to assess their risk of developing cardiovascular disease.

DETAILED DESCRIPTION:
Patients who experience a medical event are often motivated to improve their health by engaging in healthy lifestyle behaviors, such as improving their diet and beginning to exercise. For example, patients who are considered smokers prior to surgery may sometimes stop smoking following surgery. However, we are unsure of other changes following surgery. For example, we are unsure if surgery can initiate any changes in exercise and diet, and we are unsure if these changes can influence the risk of developing cardiovascular disease. Consistent and positive lifestyle changes will likely reduce an individual's risk of developing cardiovascular disease in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 - 75 years
* Scheduled for intermediate- to high risk non-cardiac surgery (intra-thoracic or intra-abdominal surgery, all vascular surgery, intra-cranial neurosurgery, spine surgery)
* Expected post-operative length of stay of at least two days, according to the surgeon's expectation
* At least two of the following CVD risk factors:

History of: Hypertension, Diabetes, Coronary artery disease, Chronic heart failure, Chronic kidney disease, Cerebrovascular disease, Peripheral vascular disease.

Obesity (BMI >25 kg/m2), Current smoking, Poor exercise capacity (<4 METS)

Exclusion Criteria:

* Currently participating in a CVD risk reduction program
* Patient is scheduled to undergo transplant or has undergone emergency surgery
* Life expectancy <1 year (palliative surgery)
* Recent (<6 months) myocardial infarction or stroke
* Surgery scheduled <1 month
* Inability to effectively communicate

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-cardiac surgery patients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Baseline assessment for calculating the pre-operative 10-year CVD event risk | 1 month before surgery
  For the baseline assessment, the expected 10-year CVD event risk of each participant will be calculated according to the appropriate CVD event risk prediction score using blood tests, questionnaire to estimate an individual's functional capacity, blood pressure, heart rate and ECG.
Follow-up assessment for calculating the post-operative 10-year CVD event risk | 3 months after surgery
  For the follow-up assessment, the expected 10-year CVD event risk of each participant will be calculated according to the appropriate CVD event risk prediction score using blood tests, questionnaire to estimate an individual's functional capacity, blood pressure, heart rate and ECG.

SECONDARY OUTCOMES:
Occurrence of Cardiovascular or Non-Cardiovascular event | 30 days after surgery
  Cardiovascular related (e.g. Myocardial infarction/injury, mortality, heart failure) or non-cardiovascular related (e.g. surgical site infections, unexpected critical care unit admissions, re-operations).

CONTACTS AND LOCATIONS:
Overall Officials: Wilton van Klei, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada